CLINICAL TRIAL: NCT01081080
Title: PITT0110 - Cardiac Magnetic Resonance: A Parallel Protocol to Cardiac Outcome Measures in Children With Muscular Dystrophy
Brief Title: Cardiac Magnetic Resonance in Children With Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Dr. Paula R. Clemens, University of Pittsburgh
Other Study IDs: PITT0110
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Duchenne Muscular Dystrophy; Becker Muscular Dystrophy; Limb Girdle Muscular Dystrophy
Keywords: cardiac; muscle; pediatric; dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This protocol will exploit novel state of the art cardiovascular magnetic resonance techniques to examine important changes in the heart in children with muscular dystrophy. The purpose of this study is to compare cardiac magnetic resonance (CMR) with the collected cardiac outcome data obtained in protocol: PITT1109 - Cardiac Outcome Measures in Children with Muscular Dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Participant enrolled in the CINRG study: PITT1109 - Cardiac Outcome Measures in Children with Muscular Dystrophy

Exclusion Criteria:

* Pregnant woman (when uncertain, participants will undergo urine testing) or lactating women
* Decompensated congestive heart failure (unable to lie flat during CMR)
* Impaired renal excretory function (calculated Glomerular Filtration Rate less than 30mL/min)
* Contra-indications to Magnetic Resonance Imaging:

  * Cardiac pacemaker or implantable defibrillator
  * Cerebral aneurysm clip
  * Neural stimulator
  * Metallic ocular foreign body
  * Harrington-rod
  * Any implanted device (i.e. insulin pump, drug infusion device)
  * Claustrophobia
  * Metal shrapnel or bullet

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from the parallel protocol: PITT1109 Cardiac Outcome Measures in Children with Muscular Dystrophy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, MD, Study Chair — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Pittsburgh, Pittsburgh, Pennsylvania